CLINICAL TRIAL: NCT06349343
Title: Clinical Study of the Safety and Efficacy of CD19/BCMA CAR-T Cell Therapy for Refractory/Moderate-to-severe Systemic Lupus Erythematosus
Brief Title: CD19/BCMA CAR-T Cell Therapy for Refractory/Moderate-to-severe Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230949
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Refractory/Moderate-to-severe systemic lupus erythematosus; CAR-T cell therapy; CD19; BCMA
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/BCMA CAR-T cell therapy intervention (Experimental): The first 3 participants will be enrolled to receive CAR-T cell infusion without pretreatment chemotherapy. Then participants' peripheral blood samples would be collected for CAR-T cell testing. If test results showed the presence of CAR-T cells on certain time points, CAR-T cell therapy without pretreatment chemotherapy is considered feasible, and the subsequent 17 participants will receive the consistent regimen; Otherwise, the 3 participants will be re-treated with pretreatment chemotherapy and CAR-T cell infusion, and the subsequent 17 participants will receive pretreatment chemotherapy-containing regimen.
  Interventions: Biological: CD19/BCMA CAR-T cell therapy

INTERVENTIONS:
Biological: CD19/BCMA CAR-T cell therapy — CD19/BCMA CAR-T cell will be infused intravenously at 3 doses: Dose A, Dose B, Dose C.

SUMMARY:
The purpose of the study is to explore the safety and efficacy of cluster of differentiation 19 (CD19)/B cell maturation antigen (BCMA) CAR-T cell therapy in refractory/moderate-to-severe systemic lupus erythematosus(SLE).

DETAILED DESCRIPTION:
The prognosis of patients with refractory/moderate-to-severe systemic lupus erythematosus (SLE) remains poor, due to two major therapeutic obstacles: (1) current treatment strategies including glucocorticoids, immunosuppressive agents, biological agents, are still difficult to achieve disease control, making the disease condition of some patients continue to be active or even worse; (2) some patients are unable to wean themselves off glucocorticoid and face the risk of numerous adverse effects caused by long-term glucocorticoid dependence, such as glucocorticoid-related diabetes, femoral head necrosis, hypertension, stress ulcers, and infection, etc. Therefore, there is a strong unmet clinical need for more effective treatment for patients suffering from refractory/moderate-to-severe SLE. Several preclinical and clinical studies have shown the efficacy of chimeric antigen receptor T (CAR-T) cell therapy in SLE. The aim of this study is to investigate the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of cluster of differentiation 19 (CD19)/B cell maturation antigen (BCMA) CAR-T cell therapy in refractory/moderate-to-severe SLE. Patients with refractory/moderate-to-severe SLE will be invited to participate in the study, to receive CD19/BCMA CAR-T cell intravenous infusion and follow-up visits of up to 1 years after enrollment. Given that the pretreatment chemotherapy (fludarabine,cyclophosphamide) of CAR-T therapy in current SLE clinical studies is mostly based on experiences in hematologic malignancies, which may cause severe complications such as infection, there is a lack of evidence-based rationale for patients with SLE to receive pretreatment chemotherapy. This study will explore the feasibility of CAR-T cell therapy without pretreatment chemotherapy in the treatment of refractory/moderate-to-severe systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Participants or their legal guardians understand and voluntarily sign the informed consent form, and be able to complete all the documents, procedures, follow-up examinations and treatments specified in the study protocol, with good compliance;
2. Age range from 18 to 70 years old, regardless of gender;
3. Participants diagnosed with SLE according to the 2019 European League Against Rheumatism (EULAR)/the American College of Rheumatology (ACR) SLE criteria at least 24 weeks prior to screening;
4. Refractory/moderate-to-severe SLE needs to meet the following criteria at screening: SELENA-SLEDAI score > 6 points; PGA ≥ 1 points; BILAG-2004 organ system scores of at least 1 A or 2 B;Have received at least 12 weeks of standardized treatment for SLE prior to screening but lack efficacy;
5. Participants with fertility agree to take effective contraceptive measures throughout the study and within 3 months after the last follow-up visit.

Exclusion Criteria:

1. Diagnosis of active severe lupus nephritis within 8 weeks prior to screening, requiring medications prohibited by the research protocol for active nephritis, hemodialysis or prednisone ≥ 100 mg/d, or equivalent glucocorticoid therapy for ≥14 days;
2. Any attempted suicide or suicidal ideation within the past year prior to screening;
3. Presence of SLE or non-SLE related central nervous system diseases or pathological changes within 8 weeks prior to screening;
4. Previous or current diagnosis of non-SLE-related inflammatory arthropathy or skin diseases;
5. History of vital organ transplantation or hematopoietic stem cell/or bone marrow transplantation;
6. History of lymphoproliferative diseases;
7. Subjects with malignancy within 5 years prior to screening;
8. Have received plasma exchange, plasma separation, hemodialysis, or intravenous immunoglobulin (IVIG) within 14 days prior to screening;
9. Other autoimmune diseases requiring systemic therapy;
10. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the lower limit of research institution's test range. Subjects with positive hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, or syphilis;
11. Active or latent tuberculosis at screening;
12. Abnormalities in major organ function at screening;
13. Previous or current diagnosis of acute or chronic illnesses unrelated to SLE with obviously unstable or uncontrollable clinical symptoms;
14. Severe lupus lung damage at screening;
15. Severe lupus cardiac damage at screening;
16. Presence of uncontrollable infections at screening, requiring antibiotic therapy;
17. Have received live/attenuated vaccination within 4 weeks prior to screening or plan to receive live/attenuated vaccination throughout the study;
18. Have received intra-articular, intramuscular or intravenous glucocorticoids within 4 weeks prior to screening;
19. Have received any commercially available Janus kinase (JAK) inhibitor or Bruton tyrosine kinase (BTK) inhibitor within 12 weeks prior to screening;
20. Have received B-cell targeted therapy prior to screening;
21. Have received a biologic agent other than B-cell targeted therapy within 5 half-lives prior to screening;
22. Previously received therapies with CAR-T cells or other genetically modified T cells;
23. Have received therapeutic dose of corticosteroids within 7 days prior to leukapheresis or within 72 hours prior to infusion;
24. Subjects that have donated blood for ≥ 400mL or had a significant blood loss equivalent to at least 400mL within 4 weeks prior to screening, or have received blood transfusion within 8 weeks, or plan to donate blood during the study period;
25. History of ≥grade 2 bleeding within 4 weeks prior to screening or need for long-term continuous anticoagulant therapy;
26. Subjects that have undergone any major surgeries within 12 weeks prior to screening, or those who are scheduled to undergo major surgery during the study period;
27. History of drug abuse within 12 weeks prior to screening;
28. Female subjects who are pregnant or lactating, or intend to conceive within 2 years after the cell infusion; male patients whose female partners intend to conceive within 2 years after the cell infusion;
29. History of any significant drug allergy or intolerance;
30. Subjects that have participated in other clinical trials within 3 months prior to screening and/or currently participated in other clinical trials (those who do not receive study drugs are excluded);
31. Presence of other circumstances that make the subjects not eligible for participation in the study, in the opinion of the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Within 1 years after CAR-T cell infusion
  Safety and tolerability will be assessed by incidence and severity of adverse events (AEs) and serious AEs (SAEs). Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) are graded by ASTCT criteria, other AEs are assessed by CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Proportion of subjects with SRI-4 response | Within 1 years after CAR-T cell infusion(month 1, month 3, month 6, month 9, month 12）
  SRI-4 response is defined as: 1) the Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score decrease by no less than 4 points from baseline; 2) the British Isles Lupus Assessment Group (BILAG) score with no new A domain score and no more than 1 new B domain score compared to baseline; 3) the Physician Global Assessment (PGA) score increase less than 0.3 point from baseline.
Changes in the Safety of Estrogens in Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score from baseline | Within 1 years after CAR-T cell infusion(month 1, month 3, month 6, month 9, month 12）
  Range [0, 105]，higher score represents worse disease activity
Changes in the BILAG-2004 score from baseline | Within 1 years after CAR-T cell infusion(month 1, month 3, month 6, month 9, month 12）
  Range [0, 72]，higher score represents worse disease activity
Changes in the Physician Global Assessment (PGA) score from baseline | Within 1 years after CAR-T cell infusion(month 1, month 3, month 6, month 9, month 12）
  Range [0, 3]，higher score represents worse disease activity
Pharmacokinetics (PK) | Within 1 years after CAR-T cell infusion(per 3 days in month 1, per month in month 2 - month 12）
  Concentration of CAR-T cell in peripheral blood will be evaluated
Pharmacodynamics (PD) | Within 1 years after CAR-T cell infusion(per 3 days in month 1, per month in month 2 - month 12）
  Pharmacodynamics (PD) will be assessed by levels of cytokines(IL-2、IL-6、IL-10、IFN-γ), changes of lymphocyte subsets, immunological indexes(IgG、IgM、IgA、IgE) in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College HUAZHONG University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No